CLINICAL TRIAL: NCT00813241
Title: A Pilot, Open-Label, Randomized, Crossover, Pharmacokinetic Study Of Enhanced Bioavailability Formulations Of Celecoxib In Healthy Volunteers
Brief Title: A Pilot Open-Label Crossover Bioavailability Study of Celecoxib in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A3191354
Record Dates: First submitted 2008-12-22; First posted 2008-12-23 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Healthy Volunteers
Keywords: Ankylosing spondylitis,Rheumatoid Arthritis,Adenomatous Polyposis Coli,Osteoarthritis,Dysmenorrhoea,pharmacokinetic study
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Active Comparator): A single dose of 200 mg celecoxib capsule administered as 1 x 200 mg celecoxib capsule, (Reference Formulation)
  Interventions: Drug: celecoxib reference formulation
- B (Experimental): A single dose of 150 mg celecoxib administered as 1 x 150 mg tablet formulation containing granule type A1
  Interventions: Drug: celecoxib test formulation A1
- C (Experimental): A single dose of 150 mg celecoxib administered as 1 x 150 mg tablet containing granule type B2
  Interventions: Drug: celecoxib test formulation B2
- D (Experimental): A single dose of 150 mg celecoxib administered as 1 x 150 mg tablet containing granule type C1
  Interventions: Drug: celecoxib test formulation C1

INTERVENTIONS:
Drug: celecoxib reference formulation — 200 mg single oral dose of celecoxib tablets
  Arms: A
Drug: celecoxib test formulation A1 — 150 mg single oral dose of celecoxib A1 formulation tablets
  Arms: B
Drug: celecoxib test formulation B2 — 150 mg single oral dose of celecoxib B2 formulation tablets
  Arms: C
Drug: celecoxib test formulation C1 — 150 mg single oral dose of celecoxib Cl formulation tablets
  Arms: D

SUMMARY:
A pharmacokinetic study in healthy volunteers to determine the relative bioavailability of three formulations of celecoxib to the approved formulation.

DETAILED DESCRIPTION:
Pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years, inclusive (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure (BP) and pulse rate measurement, 12-lead ECG and clinical laboratory tests);
* Body Mass Index (BMI) of approximately 18 to 32 kg/m2; and a total body weight >50 kg (110 lbs). A BMI lower limit of 17.5kg/m2 may be rounded up to 18.0 kg/m2, a BMI upper limit of 32.5 kg/m2 may be rounded down to 32.0 kg/m2 and will be acceptable for inclusion;
* Evidence of a personally signed and dated informed consent document indicating that the subject (or a legally acceptable representative) has been informed of all pertinent aspects of the trial;
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing);
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen;
* History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor), within 6 months of screening;
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day;
* Treatment with an investigational drug within 30 days or 5 half-lives preceding the first dose of study medication;
* 12-lead ECG demonstrating QTc >450 msec at Screening. If QTc exceeds 450 msec, the ECG should be repeated two more times and the average of the three QTc values should be used to determine the subject's eligibility;
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of non-hormonal contraception, as outlined in this protocol, from at least 14 days prior to the first dose of study medication until completion of follow-up procedures;
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication. Herbal supplements and hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) and hormone replacement therapy must be discontinued 28 days prior to the first dose of study medication. Depo-Provera® must be discontinued at least 6 months prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of less than or equal to 1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor;
* Use of grapefruit containing products within at least 7 days prior to the administration of study medication;
* Blood donation of approximately 1 pint (500 mL) within 56 days prior to dosing;
* History of sensitivity to heparin or heparin-induced thrombocytopenia;
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol;
* Subjects who have pre-existing asthma, a known hypersensitivity to celecoxib, or have experienced asthma, urticaria or allergic-type reactions after taking sulfonamides, aspirin, selective COX-2 inhibitors, or other non-steroidal anti-inflammatory drugs (NSAIDs);
* Subjects with a prior history of ulcer disease or gastrointestinal bleeding;
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
PK endpoints will include Cmax, C12h, Tmax, AUCtlqc, AUCinf, and half-life (t1/2) for each formulation as data permit | 2 months
Visual inspection of median plasma concentration versus time profiles resulting from each formulation | 2 months

SECONDARY OUTCOMES:
Adverse events and safety laboratory tests | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191354&StudyName=A%20Pilot%20Open-Label%20Crossover%20Bioavailability%20Study%20of%20Celecoxib%20in%20Healthy%20Volunteers